CLINICAL TRIAL: NCT02307786
Title: Long Term Outcomes in β Thalassemia Major - Comparing Late Outcomes Following Allogeneic Hematopoietic Stem Cell Transplantation and Standard Supportive Care
Brief Title: Long Term Outcomes in β Thalassemia Major
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: SCT 0414B
Record Dates: First submitted 2014-09-19; First posted 2014-12-04 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Beta-Thalassemiall -Transplantation
- Beta-Thalassemia Supportive Care

SUMMARY:
Beta thalassemia (β-thalassemia) is the most common genetic disease worldwide. Individuals with thalassemia are born with a defect in hemoglobin. Hemoglobin is a protein in red blood cells that carries oxygen to vital organs such as the brain, heart, lungs and kidneys. Thalassemia major is a hereditary anemia characterized by little or no ß-globin production, which results in hemolysis (breakdown or destruction of red blood cells) due to the formation of unstable alpha-globin tetramers and ineffective erythropoiesis which is uniformly fatal in the absence of regular transfusions. Although improvements in conservative treatment have improved the prognosis of thalassemia considerably disease and transfusion related complications in affected patients progress over time, causing severe morbidity and shortened life expectancy. Substantial lifelong health care expenses are also involved, often a financial burden for families and unsustainable in most developing countries.

The hypothesis is that patients who had beta thalassemia who have undergone a hematopoietic stem cell transplant (HSCT) and are >1 year post-HSCT will have less long term comorbidities and a higher quality of life (QOL) as compared to those with beta thalassemia who are maintained on supportive care. In order to assess quality of life, a quality of life questionnaire will be asked. Extraction of data from the patient's medical record will also be used to determine any comorbidities that have occurred after either a HSCT or supportive care therapy.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is considered a suitable alternative to conservative management which includes chronic transfusion therapy, iron chelation (iron overload) and management of complications of transfusion therapy and iron overload. Barriers to HSCT considerations include risks inherent to transplant- early mortality, graft versus host disease (GVHD), graft rejection, infections prior to immune reconstitution, and transplant related organ toxicities. As in supportive care, significant progress has been made in HSCT for thalassemia has been made over the last 3 decades. This has resulted in disease-free survival (DFS) rates exceeding 80% especially in young, low-risk patients with histocompatible (same gene) family donors and more recently even in unrelated donor transplants following streamlining of preparative regimen and improvements in post-HSCT supportive care.

Lucarelli and his colleagues at Pesaro initially pioneered HSCT in thalassemia and described a standard "Pesaro" risk stratification scheme based on liver size by physical examination, fibrosis detected on liver biopsy, and chelation history. This has been used for years to risk stratify patients before HSCT and has been shown to correlate well with immediate transplantation outcomes. More recently reports from the Center for International Blood and Marrow Transplant Research (CIBMTR) and from the Asian sub-continent on results of Human Leukocyte Antigen (HLA) -matched sibling HSCT for thalassemia major confirmed that age at transplantation and liver size are independent predictors of mortality after transplantation. In patients aged <7 years and without hepatomegaly (liver palpated <2 cm below the costal margin), the 5-year probabilities of Overall Survival (OS) and DFS were 98% and 94%, respectively (ref). Morbidity in thalassemia patients (both transplant related and non-transplanted) is attributed to iron overload associated end organ damage. Although there is data on long term outcomes in chronically transfused thalassemia patients, the data on long-term outcomes after HSCT for thalassemia remains limited.

Some patients undergo hematopoietic stem cell transplantation (HSCT) in hopes to cure themselves of Beta-Thalassemia. Other patients manage their Beta-Thalassemia with supportive care including chronic blood transfusions, iron chelation and medications. The purpose of this study is to compare how patients with Beta-Thalassemia are doing after HSCT versus those patients who manage their Beta-Thalassemia with supportive care. This proposal aims to compare long term outcomes in thalassemia patients that have survived a HSCT for thalassemia and compare it with the age and sex matched patients who have remained on transfusion therapy with regular chelation. In order to compare these two subsets of patients, data will be obtained from the Thalassemia Longitudinal Cohort (TLC) study.

ELIGIBILITY:
Inclusion for those who underwent HSCT:

* Age 0 to 30 years of age
* >1 year post-allogeneic HSCT for Beta-Thalassemia. Any donor (sibling or unrelated) and any donor source (bone marrow, peripheral blood, umbilical cord blood) is considered eligible. Any conditioning regimen is considered acceptable for enrollment

Exclusion:

* <1 year post-allogeneic HSCT for Beta-Thalassemia
* Patient expired prior to 1 year post-HSCT
* Autologous stem cell transplantation for Beta-Thalassemia

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will be divided into the following groups:
  * Recipients that are >1 year post allogeneic HSCT from any donor
  * Patients ('Controls') enrolled on the Thalassemia Longitudinal Cohort study and/or the Thalassemia Clinical Registry Network (TCRN) and continue to receive supportive care
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11-13 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Beta-Thalassemia patients and Quality of Life after HSCT versus supportive care therapy | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States